CLINICAL TRIAL: NCT01140854
Title: Cognitive Dysfunction in Hypertensive Patients Having Spine Surgery
Acronym: HTN
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Eric J. Heyer, MD, PhD, Professor of Anesthesiology, Clinical Operations, Columbia University
Other Study IDs: AAAD3838
Record Dates: First submitted 2010-06-02; First posted 2010-06-10 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Hypertension
Keywords: hypertension; hypotension; cognitive; neurocognitive; cognitive dysfunction; postoperative cognitive dysfunction (POCD); neuropsychometric
MeSH Terms: conditions — Hypertension; Hypotension; Cognitive Dysfunction; Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hypertension (case): Elderly patients 60 years old or older undergoing simple lumbar spine surgery under general anesthesia will receive neurologic/neuropsychometric examinations.
  Interventions: Procedure: Lumbar spine surgery; Other: Neurologic/neuropsychometric examinations
- Normotension (control): Middle-aged patients (40-60 years) undergoing simple lumbar spine surgery under general anesthesia as controls to compare their performance to those patients >60 years - will also receive neurologic/neuropsychometric examinations.
  Interventions: Procedure: Lumbar spine surgery; Other: Neurologic/neuropsychometric examinations

INTERVENTIONS:
Procedure: Lumbar spine surgery — (non-experimental) we do not intend to change the criteria of selection for simple lumbar spine surgery, anesthesia, or the postoperative management of the patients studied.
Other: Neurologic/neuropsychometric examinations — To measure postoperative cognitive dysfunction.

SUMMARY:
While hypotension during general anesthesia has routinely been considered to be a tolerable abnormality with little clinical consequence, the proposed study takes the innovative approach of defining hypotensive events within the construct of a patient's own hypertensive status, fractional mean arterial blood pressure (fMAP). Because the investigators primary variable is within the control of anesthesia personnel, the study portends a potentially simple and easy to implement treatment. The introduction of neuropsychometric measures as the relevant evaluator of post-operative cognitive dysfunction is innovative, and may be more relevant to the average elderly patient than simple mortality.

DETAILED DESCRIPTION:
After major non-cardiac and non-cerebral surgery, postoperative cognitive dysfunction (POCD) occurs in a significant percentage of patients. The consequences of POCD are profound. Elderly patients having POCD at 1 week have an increased risk of disability or voluntary early retirement, and patients having POCD at 3 months have increased mortality.

The effect of low arterial blood pressure, called hypotension, during surgery on the incidence of POCD is not obvious. This effect has been obscured in a number of previous studies because, it was assumed that hypotension had to persist for minutes to hours to be deleterious, when, in fact, the duration is uncertain. In addition, patient outcomes were not analyzed as a function of a history of hypertension. In this research application, the investigators focus specifically on patients with a history of hypertension because their physiology is different than patients with normal arterial blood pressure. These hypertensive patients may be unable to compensate for low arterial blood pressure by a process called cerebral autoregulation. As a result, patients with a history of hypertension may be at greater risk for decreased cerebral perfusion and cerebral ischemia secondary to decreased systemic arterial blood pressure even during surgery for procedures not thought to put the brain at risk of ischemia.

In a prior retrospective study, the investigators analyzed hemodynamic data from fifty elderly (average age >60 years) patients having simple lumbar spine surgery, which is not thought to be associated with cerebral ischemia. These patients were all examined with a battery of neuropsychometric tests before and after surgery. Patients with a history of hypertension had cognitive changes that are dependent on the lowest fractional mean arterial blood pressure (fMAP), where fMAP is mean arterial blood pressure (MAP) divided by baseline MAP. Such changes were not found in patients without a history of hypertension. This relationship did not depend on the steady state fMAP or the highest fMAP reached in either group.

To confirm and extend these results the investigators therefore propose and hypothesize that: In patients with a history of hypertension, compared to patients without this history, low fMAPs during induction predict cognitive performance after surgery.

To evaluate these hypotheses the investigators will determine the incidence of post-operative cognitive dysfunction (POCD) as a function of the fMAP in hypertensive and normotensive patients undergoing elective simple lumbar spine surgery.

If the proposed study demonstrates that acute intra-operative episodes of hypotension are deleterious to cognitive performance in patients with hypertension, and that there are demonstrable consequences in terms of QOL measures, the possibility of a direct and low cost intervention will be available that will lead directly to an efficacy trial using non-invasive measures of cerebral blood flow algorithms to prevent POCD.

The investigators plan to conduct a multicenter study in which 200 elderly patients (>60 years) are tested with a validated battery of 6 neuropsychometric tests before simple elective lumbar spine surgery (microdiscectomy or 1-2 level laminectomies without fusions lasting <5 hours and not requiring blood transfusions) and two times after surgery, at 24 hours and at 1 month. Two questionnaires for QOL will be performed before surgery and at 1 month. Patients will be questioned whether they have a history of hypertension, and, if they do, then its duration and treatment.

Our analysis will be based on comparing the fMAP to the neuropsychometric performance before and after surgery. To see if neuropsychometric changes occur as a component of a routine anesthetic, anesthesiologists will not be given a specific protocol for intraoperative management.

The primary outcome measure will be changes in test performance between baseline and the post-operative period at 1 day and 1 month. This primary measure will be a rating of overall change in performance compared to three values of fMAPs: lowest, steady state and highest fMAP attained. Our analysis will also include uni- and multi-variate analyses which will include and QOL.

ELIGIBILITY:
Inclusion Criteria:

* elective spine surgery
* > 60 years old
* < 5 hours of surgery
* microdiskectomy
* 1-2 levels of spinal laminectomies

Exclusion Criteria:

* transfusions
* > 5 hours of surgery
* > 2 levels of laminectomies
* spinal instrumentation

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients >60 years old will be recruited who are scheduled for elective simple spine surgery (microdiskectomy or 1-2 level laminectomies without fusion) and lasting <5 hours without blood transfusion.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Neuropsychometric changes at 1 day | Baseline to 1 Day
  The investigators will determine whether there are neuropsychometric changes associated with simple spine surgery as a function of arterial blood pressure measurements relative to the patient's baseline values at 1 day.

SECONDARY OUTCOMES:
Neuropsychometric changes at 1 Month | Baseline to 1 Month
  The investigators will determine whether there are neuropsychometric changes associated with simple spine surgery as a function of arterial blood pressure measurements relative to the patient's baseline values at 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Heyer, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Result] Yocum GT, Gaudet JG, Teverbaugh LA, Quest DO, McCormick PC, Connolly ES Jr, Heyer EJ. Neurocognitive performance in hypertensive patients after spine surgery. Anesthesiology. 2009 Feb;110(2):254-61. doi: 10.1097/ALN.0b013e3181942c7a. PMID 19194152